CLINICAL TRIAL: NCT06564636
Title: A Multi-Centre Study in Patients Undergoing Total Hip Arthroplasty With the Smith+Nephew CATALYSTEM™ Primary Hip System
Acronym: CATALYSTEM
Status: Enrolling by invitation | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CATALYST.2023.02
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-03

CONDITIONS: Total Hip Arthroplasty (THA); Osteoarthritis; Degenerative Joint Disease; Inflammatory Arthritis; Avascular Necrosis; Post-traumatic Arthritis; Congenital Hip Dysplasia
Keywords: Total Hip Arthroplasty; THA; Hip System; Hip; CATALYSTEM; CATALYST; Collared; Collarless; Cementless; Primary THA
MeSH Terms: conditions — Osteoarthritis; Joint Diseases; Arthritis; Osteonecrosis; Hip Dislocation, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CATALYSTEM: Participants who have already received or are due to receive the CATALYSTEM Cementless Primary Hip System
  Interventions: Device: CATALYSTEM

INTERVENTIONS:
Device: CATALYSTEM — CATALYSTEM Cementless Primary Hip System for participants with Total Hip Arthroplasty

SUMMARY:
A Multi-Center Study in Patients Undergoing Total Hip Arthroplasty with the Smith+Nephew CATALYSTEM™ Primary Hip System. The purpose of the study is to assess safety and performance of the CATALYSTEM™ and to support product approval in global markets.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, non-randomized study of subjects implanted with the CATALYSTEM™ Primary Hip System for primary Total Hip Arthroplasty (THA). Subjects will be enrolled and followed for 5 years post-operatively to assess safety and efficacy of the CATALYSTEM™ Primary Hip System. The primary objective is to assess 2-year post-operative stem survivorship of the CATALYSTEM™ Hip System (i.e. the femoral stem with all its variants and instrumentation) in primary THA procedures for each stem type (Collared/Collarless). Stem survivorship is defined as no aseptic revision of the implanted femoral stem.

ELIGIBILITY:
Inclusion Criteria:

1. a. Subject needing primary THA due to end stage degenerative joint disease (primary diagnosis of osteoarthritis), avascular necrosis, post-traumatic arthritis, inflammatory arthritis, or congenital hip dysplasia.

OR

1. b. Subject has undergone primary THA with the S+N CATALYSTEM™ Primary Hip stem in the past 12 months for end stage degenerative joint disease (primary diagnosis of osteoarthritis), avascular necrosis, post-traumatic arthritis, inflammatory arthritis, or congenital hip dysplasia and all the following conditions have been met for the appropriate timepoint:

   * Preoperative Patient Reported Outcome Measures (PROMs):

     * Hip Disability and Osteoarthritis Outcome Score Junior (HOOS, JR.)
     * European Quality of Life (EuroQol) Five-dimensional Five-level (EQ-5D-5L), and
   * Radiographs have been obtained:

     ° Anterior Posterior (AP) Pelvis
     * AP Hip*, and
     * Lateral**
   * 6-Weeks

     ° PROMs (HOOS, JR., and EQ-5D-5L), and
     * Radiographs (AP Pelvis, AP Hip*, and Lateral**) have been obtained or these can be collected prospectively in window per schedule of events, and
   * 1-Year

     ° PROMs (HOOS, JR., and EQ-5D-5L), and

     ° Radiographs (AP Pelvis, AP Hip*, and Lateral**) have been obtained or these can be collected prospectively in window per schedule of events

     2. Subject agrees to consent and to follow the prospective study visit schedule by signing the Independent Review Board (IRB)/Independent Ethics Committee (IEC) approved Informed Consent Form (ICF).

     3. Subject is eighteen to eighty (18-80) years old (inclusive).

     4. Subject can read, understand, and communicate responses to the PROMs.

footnote:

*For the AP Hip radiograph, sites MUST ensure that positioning (standing AP Hip vs. supine AP Hip) is consistent across all study visits for an individual subject (i.e. if subject had standing AP Hip at pre-op then collect standing AP Hip at all visits for that subject).

** Lateral radiograph is to include any one of the following, but for standardization, sites MUST ensure consistency across all study visits for an individual subject: Cross-Table Lateral (CTL) or Frog-lateral or lateral femoral/Lowenstein (i.e. if subject had frog-leg lateral at pre- op then collect frog-leg lateral at all visits for that subject).

Exclusion Criteria: Any one (1) of the following criteria will disqualify a potential subject from participation in the study:

1. Subject has conditions that would eliminate or tend to eliminate adequate implant support or prevent the use of an appropriately-sized implant, e.g.:

   * Blood supply limitations
   * Insufficient quantity or quality of bone support e.g., osteoporosis, or metabolic disorders which may impair bone formation, and or osteomalacia
   * Mental or neurological conditions which may tend to impair the patient's ability or willingness to restrict activities; or impairing or precluding cooperation with post-operative protocols including mental illness, drug or alcohol abuse.
   * Physical conditions or activities which tend to place extreme loads on implants and may impair short and long-term satisfactory results of the implant, e.g., Charcot joints, muscle deficiencies, multiple joint disabilities, etc.
   * Infections or other conditions which may lead to increased bone resorption
   * Skeletal immaturity
2. Subject has a Body Mass Index (BMI) >/= 45 at time of surgery.
3. Subject has a known allergy to one or more components of the study device.
4. Any subject that meets the definition of a Vulnerable Subject per ISO 14155 Section 3.55 (i.e., individuals who are unable to fully understand all aspects of the investigation that are relevant to the decision to participate, or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response).
5. Subject is entered in another drug, biologic, or device study or has been treated with an investigational product 30 days prior to the surgery date.
6. Subject is known to be at risk for lost to follow-up, or failure to return for scheduled visits.
7. Women who are pregnant or nursing.
8. Subject has participated previously in this clinical trial and has been withdrawn.
9. Subject has an active infection - systemic or at the site of intended surgery.
10. Subject had a contralateral (opposite) hip replacement that was implanted less than 3 months prior to consent, is scheduled for a simultaneous contralateral hip implant, or plans to have their contralateral hip implanted within 3 months following this study-specific implant (known as 'staged bilateral THA').
11. Subject with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who meet the inclusion and exclusion criteria at participating sites in both the United States and Canada.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
CATALYSTEM™ femoral stem implant survivorship 2 years post-operatively by stem type (collared/collarless) | 2 years post-operative
  Stem survivorship is defined as no aseptic revision of the implanted femoral stem

SECONDARY OUTCOMES:
CATALYSTEM™ femoral stem implant survivorship rates by stem type (collard/collarless) | 6 weeks, 1 year, and 5 years post-operative
  Implant survivorship is defined as no aseptic stem revision
Hip Disability and Osteoarthritis Outcome Score, Junior (HOOS Jr) | Pre-operative, 6 weeks, 1 year, 2 years, and 5 years post-operative
  Patient-administered self-report survey based on the HOOS that specifically focuses on the outcome after THA. HOOS, JR. consists of 2 areas: pain (2 items) and function, daily living (4 items). The last week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes - none, mild, moderate, severe, extreme) and each question gets a score from 0 to 4. An interval score from 0 -100 (0 indicating total hip disability and 100 indicating perfect hip health) is calculated.
EuroQol 5-Dimension 5-Level Visual Analogue Scale (EQ-5D-5L VAS) | Pre-operative, 6 weeks, 1 year, 2 years, and 5 years post-operative
  The VAS records the subject's self-rated health on a vertical visual analogue scale. The endpoints on the scale are labelled "The best health you can imagine" and "The worst health you can imagine". Participants indicate a numerical value from 1-100 where 0 is the worst imaginable health state and 100 is the best imaginable health state. The VAS can be used as a quantitative measure of health outcome as judged by the individual respondents.
Quality of Life (EQ-5D-5L) Index Score | Pre-operative, 6 weeks, 1 year, 2 years, and 5 years post-operative
  The descriptive system is used to describe the subject's health state & consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels to choose the most appropriate answer: no problems, slight problems, moderate problems, severe problems, and extreme problems. The subject is asked to indicate his/her health state by marking the most appropriate statement in each of the five areas. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. For instance, 'slight problems' (e.g. 'I have slight problems in walking about') is always coded as '2'.) The digits for the 5 dimensions are combined in a 5-digit code. The EQ- 5D-5L index value is derived by using the vendor supplied calculator to convert each 5-digit EQ-5D-5L profile. A higher number is a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Jahnke, Study Director — Smith & Nephew, Inc.
Locations (10):
- United States (6):
  - University of California at San Francisco, San Francisco, California
  - Connecticut Orthopaedic Institute, Hamden, Connecticut
  - Orlando Health Inc., Orlando, Florida
  - Illinois Bone and Joint Institute, Des Plaines, Illinois
  - NYU Langone Health Orthopedic Hospital, New York, New York
  - Duke Health, Morrisville, North Carolina
- Canada (4):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Concordia General Hospital, Winnipeg, Manitoba
  - London Health Sciences Centre (LHSC), London, Ontario

IPD SHARING:
Plan to Share IPD: Undecided